CLINICAL TRIAL: NCT02422199
Title: A Study of Pyrotinib Plus Capecitabine Versus Lapatinib Plus Capecitabine in Patients With HER2+Metastatic Breast Cancer Who Have Prior Received Anthracyclin, Taxane or Trastuzumab
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR-BLTN-I/II-MBC
Record Dates: First submitted 2015-04-16; First posted 2015-04-21 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: HER2 Positive Metastatic Breast Cancer
MeSH Terms: interventions — pyrotinib; Lapatinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pyrotinib plus capecitabine (Experimental): pyrotinib(400 mg once daily) + capecitabine (2000 mg/m^2 daily, 1000 mg/m^2 BID)
  Interventions: Drug: pyrotinib; Drug: capecitabine
- lapatinib plus capecitabine (Active Comparator): lapatinib (1250 mg once daily) + capecitabine (2000 mg/m^2 daily, 1000 mg/m^2 BID)
  Interventions: Drug: Lapatinib; Drug: capecitabine

INTERVENTIONS:
Drug: pyrotinib
  Arms: pyrotinib plus capecitabine
Drug: Lapatinib
  Arms: lapatinib plus capecitabine
Drug: capecitabine

SUMMARY:
Pyrotinib is an oral tyrosine kinase inhibitor targeting both HER-1 and HER-2 receptors. This study is a randomized, multi-center, multinational, open-label, active-controlled, parallel design study of the combination of pyrotinib plus capecitabine versus the combination of lapatinib plus capecitabine in HER2+ MBC patients who have prior received anthracyclin, taxane or trastuzumab. Patients will be stratified by weather have prior use of trastuzumab and randomized in a 1:1 ratio to one of the following treatment arms:

* Arm A: pyrotinib (400 mg once daily) + capecitabine (1000 mg/m^2 twice daily)
* Arm B: lapatinib (1250 mg once daily) + capecitabine (1000 mg/m^2 twice daily) Patients will receive either arm of therapy until the occurrence of death, disease progression, unacceptable toxicity, or other specified withdrawal criterion.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 and ≤70 years.
* ECOG performance status of 0 to 1.
* Life expectancy of more than 12 weeks.
* At least one measurable lesion exists.(RECIST 1.1).
* Histologically or cytologic confirmed HER2 positive advanced breast cancer which failed prior therapies.
* Required laboratory values including following parameters:

ANC: ≥ 1.5 x 10^9/L;Platelet count: ≥ 100 x 10^9/L;Hemoglobin: ≥ 9.0 g/dL;Total bilirubin: ≤ 1.5 x upper limit of normal (ULN);ALT and AST: ≤ 1.5 x ULN;BUN and creatine clearance rate: ≥ 50 mL/min;LVEF: ≥ 50%;QTcF: < 470 ms for female and < 450 ms for male.

* Signed informed consent

Exclusion Criteria:

* Received previous therapy with lapatinib, neratinib, pyrotinib or any other HER2 directe tyrosine kinase inhibitor.
* Received previous therapy with capecitabine within 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-10 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Safety(adverse Events [AEs] and Serious Adverse Events [SAEs]) | : From consent through 28 days following treatment completion (estimated 18 months)
Objective Response Rate (ORR) | Estimated 12 months

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Estimated 18 months
Time to Progression (TTP) | Estimated 18 months
Duration of Response (DOR) | Estimated 18 months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - 307 Hospital Affiliated to Academy Military Medical Science, Beijing

REFERENCES:
- [Derived] Bao Y, Zhang Z, He X, Cai L, Wang X, Li X. Cost-Effectiveness of Pyrotinib Plus Capecitabine versus Lapatinib Plus Capecitabine for the Treatment of HER2-Positive Metastatic Breast Cancer in China: A Scenario Analysis of Health Insurance Coverage. Curr Oncol. 2022 Aug 23;29(9):6053-6067. doi: 10.3390/curroncol29090476. PMID 36135045